CLINICAL TRIAL: NCT05058950
Title: An Observational Study Using Multimodal Sensors to Measure Cognitive Health in Adults and Distinguish Mild Cognitive Impairment From Normal Aging
Acronym: Intuition
Status: Terminated | Type: Observational
Why Stopped: Study was terminated early as part of Biogen's ongoing research and development portfolio management efforts.
Sponsor: Biogen (Industry)
Collaborators: Apple Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 285PI401
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Mild Cognitive Impairment; Normal Aging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Phenotyped in Research Objectively: Cognitively Normal: Participants with age ≥50 years and with a label of "cognitively normal" or its equivalent based on a clinical or research evaluation in the past 24 months will be enrolled virtually.
- Phenotyped in Research Objectively: MCI: Participants with age ≥50 years, with a label of "MCI" or its equivalent based on a clinical or research evaluation in the past 24 months will be enrolled virtually.
- Phenotyped in Research Objectively: Exploratory Biomarker: Participants with age ≥50 years, with documented positive result for an Alzheimer's disease biomarker, and with a label of "subjective cognitive complaints" or "cognitively normal" or its equivalent based on a clinical or research evaluation in the past 24 months will be enrolled virtually.
- Aging Across Adulthood: MCI: Participants with age ≥50 years, with a diagnosis of MCI, mild neurocognitive disorder (MND), or cognitively impaired, not demented (CIND) will be enrolled virtually from the community.
- Aging Across Adulthood: Subjective Cognitive Complaint: Participants with age ≥50 years and positive screen result from Cognitive Function Instrument (CFI) will be enrolled virtually from the community.
- Aging Across Adulthood: Cognitively Normal With Risk Factor For Dementia: Participants with age ≥60 years and self-reported history of a minimum of 2-4 risk factors for cognitive decline will be enrolled virtually from the community.
- Aging Across Adulthood: Cognitively Normal Without Risk Factors For Dementia: Participants with age ≥60 years having missing descriptor of minimal risk factors for cognitive decline will be enrolled virtually from the community.
- Aging Across Adulthood: Cognitively Normal: Participants with age 21 to 59 years will be enrolled virtually from the community.

SUMMARY:
The primary objectives are to develop and validate a classifier using multimodal passive sensor data and metrics derived from normal iPhone and Apple Watch usage to distinguish individuals with normal cognition from those with mild cognitive impairment (MCI) and to develop and validate a cognitive wellness score that tracks fluctuations in cognitive performance over time using multimodal passive sensor data and metrics derived from normal iPhone and Apple Watch usage.

ELIGIBILITY:
Key Inclusion Criteria:

* Fluent in spoken and written English
* Minimum 8 years of education or 8th grade equivalent.
* Willing to authorize the use of confidential health information in accordance with applicable privacy regulations.
* Willing to wear an Apple Watch for daily use for the duration of the study.
* Willing to use their personal iPhone for routine daily use for the duration of the study.
* Technical requirements:

iPhone models: iPhone 8 or newer iOS versions: current publicly available iOS version

* Access to one of the following personal computing devices. Microsoft Windows based personal computers (laptops and desktops) Mac personal computers (laptops and desktops) Apple iPad tablets
* Access to WiFi or hardwired internet access in participant's place of residence.
* Active email address for enrollment account creation and for use in relaying study information.
* Active mobile telephone number for use in relaying study information when appropriate.
* Primary address within the United States (50 states and Washington, DC; not a post office (PO) box).

Key Exclusion Criteria:

* Inability to comply with study requirements.
* Any self-reported medical history of dementia (such as Alzheimer's disease, frontotemporal dementia, dementia with Lewy body, vascular dementia, rapidly progressive dementia, or Parkinson's disease dementia).
* Self-reported dependence on others to perform core activities of daily living, including feeding, dressing, bathing, toileting, or grooming.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 21 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population include participants with or without mild cognitive impairment.
Sampling Method: Non-Probability Sample
Enrollment: 22720 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the Classifier in Distinguishing Between Individuals With and Without MCI | Up to Month 23
  A classifier is a mathematical function that uses collected data to calculate the probability that an individual belongs in a given category. The reference standard for the classifier is clinical diagnosis of MCI in normal clinical care or in a research cohort.
Correlation Between the Cognitive Wellness Score and the Neuropsychological Testing Battery Score | Up to Month 23
  To develop and validate a cognitive wellness score that tracks fluctuations in cognitive performance over time using multimodal passive sensor data and metrics derived from normal iPhone and Apple Watch usage.

SECONDARY OUTCOMES:
Sensitivity and Specificity of the Classifier in Predicting Between Individuals Who Do and Do Not Develop MCI | Up to Month 23
  A classifier is a mathematical function that uses collected data to calculate the probability that an individual belongs in a given category. The reference standard for the classifier is clinical diagnosis of MCI in normal clinical care or in a research cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Virtual App-Based Study, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com
URL: https://vivli.org/

REFERENCES:
- [Derived] Butler PM, Yang J, Brown R, Hobbs M, Becker A, Penalver-Andres J, Syz P, Muller S, Cosne G, Juraver A, Song HH, Saha-Chaudhuri P, Roggen D, Scotland A, Silveira N, Demircioglu G, Gabelle A, Hughes R, Erkkinen MG, Langbaum JB, Lingler JH, Price P, Quiroz YT, Sha SJ, Sliwinski M, Porsteinsson AP, Au R, Bianchi MT, Lenyoun H, Pham H, Patel M, Belachew S. Smartwatch- and smartphone-based remote assessment of brain health and detection of mild cognitive impairment. Nat Med. 2025 Mar;31(3):829-839. doi: 10.1038/s41591-024-03475-9. Epub 2025 Mar 4. PMID 40038507
- See also: For additional information about the study: https://www.intuitionstudy.com/ — https://www.intuitionstudy.com/